CLINICAL TRIAL: NCT00113789
Title: Randomized, Phase 2 Study of Pegfilgrastim Given on the Last Day of a Multi-Day Topotecan Regimen or the Day After in Subjects With Relapsed or Refractory Ovarian Cancer
Brief Title: Evaluating Pegfilgrastim and a Multi-Day Topotecan Regimen in Subjects With Relapsed or Refractory Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 20030122
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; topotecan; neutropenia; Neulasta®
MeSH Terms: conditions — Ovarian Neoplasms; Neutropenia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Pegfilgrastim (Active Comparator)
  Interventions: Other: PI Discretion
- Placebo (Placebo Comparator)
  Interventions: Other: PI Discretion

INTERVENTIONS:
Other: PI Discretion — PI Discretion

SUMMARY:
This trial will provide data on the safety and efficacy of pegfilgrastim, in terms of duration of grade 4 neutropenia, when administered on the last day or the day after a multi-day, myelosuppressive chemotherapy regimen for ovarian cancer.

ELIGIBILITY:
Inclusion Criteria: - Subjects with histologically confirmed primary peritoneal carcinoma, epithelial ovarian cancer, or tubal carcinoma relapsed after or refractory to 1 or 2 prior regimens of therapy - Measurable or evaluable disease - GOG Performance Status of 0 to 2 - Subjects must be at least 2 weeks from major surgery and recovered from all associated toxicities or sequelae - At least 2 weeks from radiation therapy and recovered from all associated toxicities - Adequate hemopoietic function evidenced by: *ANC greater than 1.5 x 10^9/L, *platelets greater than 100 x 10^9/L and *hemoglobin greater than or equal to 10 g/dL - AST and ALT less than 1.5 x ULN; total serum bilirubin less than or equal to 2.0 mg/dL; serum creatinine less than or equal to 1.5 mg/dL or calculated creatinine clearance greater than or equal to 60 mL/min Exclusion Criteria: - Epithelial ovarian tumors of low malignant potential - Prior therapy with topotecan - Active infection requiring treatment with systemic (intravenous or oral) anti-infectives (antibiotic, antifungal, or antiviral agent) within 72 hours of chemotherapy - Prior malignancy within the last 5 years, with the exception of surgically cured basal/squamous skin cell carcinoma, and/or carcinoma of the cervix in-situ - History of impaired cardiac status (e.g., severe heart disease, cardiomyopathy, or congestive heart failure) - Any premalignant myeloid condition or any malignancy with myeloid characteristics (e.g., myelodysplastic syndromes, acute or chronic myelogenous leukemia - Subject is pregnant (e.g., positive HCG test) or breast feeding - Subject is of child-bearing potential and does not agree to using adequate contraceptive precautions - Any psychiatric, addictive or other kind of disorder which compromises the ability of the subject to give written informed consent and/or to comply with study protocol procedures - Other investigational procedures are excluded. Subject is currently enrolled in, or has not yet completed at least 30 days since ending another investigational device or drug trial(s) or is receiving other investigational agent(s)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-10; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Duration of Grade 4 Neutropenia | During treatment

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_11_GCSFSD01_20030122.pdf
- See also: FDA-approved Drug Labeling — http://www.neulasta.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com